CLINICAL TRIAL: NCT00254540
Title: Phase II Study Of Single-Agent SU011248 In The Treatment Of Patients With Renal Cell Carcinoma
Brief Title: Study of SU011248 in Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181072
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2010-02-11 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: Ph2, RCC, SU011248, SUNITINIB
MeSH Terms: conditions — Carcinoma, Renal Cell; Primary hyperoxaluria type 2 | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SU-011248 capsule (Experimental)
  Interventions: Drug: SU011248 capsule

INTERVENTIONS:
Drug: SU011248 capsule — 50mg, PO on day 28 of each 42 day cycle, until progression or unacceptable toxicity develops

SUMMARY:
To determine the objective tumor response of single-agent SU011248 at a dose of 50 mg orally once daily for 4 consecutive weeks and 2 weeks rest, repeated every 6 weeks in patients with metastatic Renal Cell Cancer (RCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma with metastases with a component of clear cell histology

Exclusion Criteria:

* Any cellular therapy (LAK, TIL, DC), any vaccine therapy, mini-transplantation, or systemic molecular-targeting therapy for RCC.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Japan (11):
  - Pfizer Investigational Site, Akita, Akita
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Tsukuba, Ibaragi
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Sayama, Osaka
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Sunto-gun, Shizuoka
  - Pfizer Investigational Site, Tokushima, Tokushima
  - Pfizer Investigational Site, Chuo-ku, Tokyo
  - Pfizer Investigational Site, Yamagata, Yamagata
  - Pfizer Investigational Site, Fukuoka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181072&StudyName=Study%20of%20SU011248%20in%20patients%20with%20advanced%20kidney%20cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- First-line Treatment Population: SU-011248 capsule:
  Subjects who had not had any prior systemic treatment for renal cell carcinoma. Subjects received SU-011248 in an open-label manner at a starting dose of 50-mg once daily for 4 consecutive weeks followed by a 2-week off-treatment period to form a complete cycle of 6 weeks. SU-011248 was taken orally in the morning without regard to meals beginning on Day 1 of the study. Subjects were monitored for toxicity, and the SU-011248 dose could be adjusted according to individual subject tolerance. Subjects were allowed to continue to receive SU-011248 until they met any of the study discontinuation criteria.
- Pretreated Population: SU-011248 capsule:
  Subjects who had previously been treated with one cytokine-based systemic therapy regimen for renal cell carcinoma. Subjects received SU-011248 in an open-label manner at a starting dose of 50-mg once daily for 4 consecutive weeks followed by a 2-week off-treatment period to form a complete cycle of 6 weeks. SU-011248 was taken orally in the morning without regard to meals beginning on Day 1 of the study. Subjects were monitored for toxicity, and the SU-011248 dose could be adjusted according to individual subject tolerance. Subjects were allowed to continue to receive SU-011248 until they met any of the study discontinuation criteria.
Period: Overall Study
Arm/Group | First-line Treatment Population | Pretreated Population
Started | 25 (All 25 subjects enrolled were included in Intent-To Treat population.) | 26 (All 26 subjects enrolled were included in Intent-To Treat population.)
Completed | 6 | 4
Not Completed | 19 | 22
Not completed — Adverse Event | 6 | 7
Not completed — Lack of Efficacy | 13 | 13
Not completed — Death | 0 | 1
Not completed — Laboratory Test Abnormality | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First-line Treatment Population | Pretreated Population | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Customized [Number; unit: participants]
  20-44 years | 4 | 1 | 5
  45-64 years | 14 | 14 | 28
  >=65 years | 7 | 11 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 11 | 21 | 32
Region of Enrollment [Number; unit: participants]
  Japan | 25 | 26 | 51
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Score 0: Fully active, able to carry on all pre-disease performance without restriction.
  Score 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  participants
    Score 0 | 20 | 22 | 42
    Score 1 | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Objective Response
Description: Based on Extramural Review Committee's assessment. Number of subjects with objective response is defined as sum of the subjects with confirmed complete response (CR) and partial response (PR) as the best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses were those that persisted on repeat imaging study ≥4 weeks after initial documentation of response. CR = the disappearance of all target lesions. PR = a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycles 1-4
Population: Intent-to-Treat (ITT) population defined as all subjects enrolled in study that receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 25 | 26
participants
  Total Number of Subjects with CR+PR | 12 | 12
  Complete Response (CR) | 1 | 0
  Partial Response (PR) | 11 | 12
Statistical Analysis 1: Comparison: First-line Treatment Population; Test type: Superiority or Other; Objective Response Rate(percentage) = 48.0, 95% CI [27.8 to 68.7]
Statistical Analysis 2: Comparison: Pretreated Population; Test type: Superiority or Other; Objective Response Rate(percentage) = 46.2, 95% CI [26.6 to 66.6]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the date of first dose of study treatment to the date of the first documentation of progressive disease (PD) or death.
Time Frame: Day 28 of Cycle 1-4, Day 28 of even cycles after Cycle 5, and at the end of the study. Up to 28 days after the last administration of the study drug.
Population: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 25 | 26
Weeks | 53.0 [3.9 to 130.0] | 46.0 [10.0 to 124.1]

3. Secondary Outcome: Time To Tumor Progression (TTP)
Description: Time to tumor progression (TTP) is defined as the time from the date of first dose of study treatment to the date of the first documentation of progressive disease (PD).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 25 | 26
Weeks | 53.0 [3.9 to 130.0] | 46.0 [10.0 to 124.1]

4. Secondary Outcome: Duration of Response (DR)
Description: Duration of response (DR) is defined as the period between the day of initial confirmation of complete response (CR) or partial response (PR) and the day of initial confirmation of progressive disease (PD) or death of any cause. For subjects who were not confirmed to have PD or death of any cause during the study (including 28 days after the completion of study treatment) or before the initiation of another antitumor therapy, DR was censored on the final confirmation of progression-free condition during the study.
Time Frame: as for outcome 2
Population: Among Intent-To-Treat population, the number of subjects with objective tumor response based on investigator's assessment was 13 and 14 for the First-line treatment and the Pretreated populations, respectively.
Measure: Median (Full Range); unit: Weeks
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 13 | 14
Weeks | 111.6 [27.1 to 111.6] | 38.1 [18.7 to 102.1]

5. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time to tumor response (TTR) is defined as the period between the day of initial study treatment and the day of initial confirmation of complete response (CR) or partial response (PR). CR = the disappearance of all target lesions. PR = a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycle 1-4, Day 28 of even cycles after Cycle 5, and at the end of the study.
Population: as for outcome 4
Measure: Median (Full Range); unit: Weeks
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 13 | 14
Weeks | 10.0 [3.6 to 34.0] | 10.5 [3.7 to 38.6]

6. Secondary Outcome: Overall Survival Time
Description: Overall survival time is defined as the time from the date of first dose of study treatment to the date of the death due to any cause. For subjects whose death had not been confirmed, overall survival time was censored on the last date when the subject was known to be alive.
Time Frame: once year. Up to 3 years after the completion of subject registration.
Population: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 25 | 26
Weeks | 143.4 [13.7 to 149.3] | 141.0 [17.0 to 141.1]

7. Secondary Outcome: Change From Baseline of European Quality of Life Questionnaire- 5 Dimensions(EQ-5D) Questionnaires Health State Index Score
Description: Change from Baseline: weighted health state index at each observation minus weighted health state index at baseline. The EQ-5D evaluates 5 dimensions of health. The subjects rates the severity of impairment for each dimensions on a 3-point scale (1 to 3). The digits for five dimensions were combined in a five-digit number describing the respondent's health state. Health states were converted into a weighted health state index (Range: 0 to 1). High score is indicating high health.
Time Frame: Day 28 of Cycle 1; Days 1 and 28 of Cycles 2-4
Population: Intent-to-Treat (ITT) population defined as all subjects enrolled in study that receive at least 1 dose of study medication.
  n=Number of subjects with analyzable data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 25 | 26
Scores on a scale
  Cycle 1 Day 28 (n=25, 24) | -0.0937 (0.2032) | -0.0604 (0.1753)
  Cycle 2 Day 1 (n=20, 23) | -0.0067 (0.1556) | 0.0513 (0.0906)
  Cycle 2 Day 28 (n=20, 22) | -0.0946 (0.2045) | -0.0957 (0.2127)
  Cycle 3 Day 1 (n=17, 21) | 0.0375 (0.1509) | 0.0153 (0.0911)
  Cycle 3 Day 28 (n=17, 21) | -0.1058 (0.2058) | -0.0735 (0.2245)
  Cycle 4 Day 1 (n=14, 19) | -0.0079 (0.1856) | 0.0173 (0.1105)
  Cycle 4 Day 28 (n=14, 21) | -0.1573 (0.1627) | -0.0974 (0.1979)

8. Secondary Outcome: Change From Baseline of European Quality of Life Questionnaire- 5 Dimensions(EQ-5D) Questionnaires Visual Analog Scale (VAS)
Description: Change from Baseline: weighted health state VAS score at each observation minus weighted health state VAS score at baseline.
  The VAS is a self-completed scale designed to rate the subject's current health state from 0 to 100 where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Day 28 of Cycle 1; Days 1 and 28 of Cycles 2-4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | First-line Treatment Population | Pretreated Population
Number analyzed (Participants) | 25 | 26
Scores on a scale
  Cycle 1 Day 28 (n=25, 24) | -11.12 (16.29) | -10.54 (15.97)
  Cycle 2 Day 1 (n=20, 23) | -2.10 (13.49) | 4.17 (13.12)
  Cycle 2 Day 28 (n=20, 22) | -7.85 (18.31) | -11.82 (24.36)
  Cycle 3 Day 1 (n=17, 21) | 2.71 (12.88) | 1.10 (9.14)
  Cycle 3 Day 28 (n=17, 21) | -12.35 (23.69) | -7.67 (18.53)
  Cycle 4 Day 1 (n=14, 19) | -1.86 (17.81) | -0.79 (19.81)
  Cycle 4 Day 28 (n=14, 21) | -11.43 (19.70) | -6.43 (19.48)

9. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-011248 in First-line Treatment Population
Description: Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration
Time Frame: Days 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 plasma concentration data for Pharmacokinetic analysis.
  n=Number of subjects with analyzable data.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | First-line Treatment Population
Number analyzed (Participants) | 25
ng/mL
  Cycle 1 Day 14 (n=24) | 81.60 (28.03) [34.30 to 163.00]
  Cycle 1 Day 28 (n=9) | 71.00 (34.23) [43.30 to 130.00]
  Cycle 2 Day 1 (n=6) | 1.24 (1.98) [0.20 to 3.85]
  Cycle 2 Day 28 (n=4) | 61.45 (17.65) [55.30 to 102.00]
  Cycle 3 Day 28 (n=4) | 71.30 (22.97) [49.70 to 84.30]

10. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-011248 in Pretreated Population
Description: Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration.
Time Frame: Days 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 plasma concentration data for Pharmacokinetic analysis.
  n=Number of subjects with analyzable data.
  Descriptive statistics on "Cycle 2 Day 1" and "Cycle 3 Day 28" were not calculated because number of subjects with analyzable data was less than 3.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Pretreated Population
Number analyzed (Participants) | 26
ng/mL
  Cycle 1 Day 14 (n=13) | 85.90 [69.90 to 119.0]
  Cycle 1 Day 28 (n=4) | 75.00 [56.60 to 151.00]
  Cycle 2 Day 28 (n=3) | 57.70 [47.00 to 61.30]

11. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-012662 in First-line Treatment Population
Description: SU-012662 is a metabolite of SU-011248. Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration
Time Frame: Days 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | First-line Treatment Population
Number analyzed (Participants) | 25
ng/mL
  Cycle 1 Day 14 (n=24) | 36.10 (20.65) [12.40 to 96.40]
  Cycle 1 Day 28 (n=9) | 50.50 (19.65) [12.70 to 66.20]
  Cycle 2 Day 1 (n=6) | 2.14 (1.21) [0.66 to 3.91]
  Cycle 2 Day 28 (n=4) | 35.15 (7.17) [21.00 to 35.70]
  Cycle 3 Day 28 (n=4) | 33.55 (13.81) [20.40 to 53.00]

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-012662 in Pretreated Population
Description: as for outcome 11
Time Frame: Days 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 plasma concentration data for Pharmacokinetic analysis.
  Descriptive statistics on "Cycle 2 Day 1" and "Cycle 3 Day 28" were not calculated because number of subjects with analyzable data was less than 3.
  n=Number of subjects with analyzable data.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Pretreated Population
Number analyzed (Participants) | 26
ng/mL
  Cycle 1 Day 14 (n=13) | 31.60 [21.10 to 57.30]
  Cycle 1 Day 28 (n=4) | 25.70 [16.10 to 39.30]
  Cycle 2 Day 28 (n=3) | 17.50 [13.90 to 29.30]

13. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-011248+SU-012662 in First-line Treatment Population
Description: SU-012662 is a metabolite of SU-011248. Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration.
  The Ctrough for total drug (SU-011248+SU-012662) was calculated as the mean of the Ctrough of total drug from each individual subject.
Time Frame: Days 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | First-line Treatment Population
Number analyzed (Participants) | 25
ng/mL
  Cycle 1 Day 14 (n=24) | 130.30 (45.31) [50.30 to 259.40]
  Cycle 1 Day 28 (n=9) | 137.20 (48.85) [63.40 to 180.50]
  Cycle 2 Day 1 (n=6) | 3.67 (2.31) [0.86 to 7.76]
  Cycle 2 Day 28 (n=4) | 93.95 (24.17) [82.40 to 136.90]
  Cycle 3 Day 28 (n=4) | 114.70 (22.83) [70.10 to 117.60]

14. Secondary Outcome: Trough Plasma Concentration (Ctrough) of SU-011248+SU-012662 in Pretreated Population
Description: SU-012662 is a metabolite of SU-011248. Trough Plasma Concentration (Ctrough) means the concentration prior to study drug administration.
  The Ctrough for total drug (SU011248+SU012662) was calculated as the mean of the Ctrough of total drug from each individual subject.
Time Frame: Days 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: as for outcome 12
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Pretreated Population
Number analyzed (Participants) | 26
ng/mL
  Cycle 1 Day 14 (n=13) | 115.10 [96.70 to 176.30]
  Cycle 1 Day 28 (n=4) | 100.70 [72.70 to 190.30]
  Cycle 2 Day 28 (n=3) | 75.20 [60.90 to 90.60]

15. Secondary Outcome: Plasma Concentrations of Vascular Endothelial Growth Factor (VEGF)
Description: Plasma concentrations of potential pharmacodynamic markers; Vascular Endothelial Growth Factor (VEGF)
Time Frame: Days 1, 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: All enrolled subjects who received at least 1 dose of study medication and who had at least 1 plasma concentration data for Pharmacodynamic analysis.
  n=Number of subjects with analyzable data.
Measure: Median (Full Range); unit: pg/mL
Groups:
- Overall: SU-011248 Capsule:First-line Treatment population plus Pretreated population
Arm/Group | Overall
Number analyzed (Participants) | 51
pg/mL
  Cycle 1 Day 1 (n=51) | 54.90 (84.99) [19.70 to 396.50]
  Cycle 1 Day 14 (n=42) | 186.60 (267.19) [60.70 to 1100.50]
  Cycle 1 Day 28 (n=16) | 259.90 (263.44) [101.00 to 977.50]
  Cycle 2 Day 1 (n=18) | 57.35 (94.18) [21.80 to 335.80]
  Cycle 2 Day 28 (n=8) | 264.75 (115.19) [120.50 to 474.90]
  Cycle 3 Day 28 (n=6) | 194.15 (111.20) [94.10 to 503.00]

16. Secondary Outcome: Plasma Concentrations of Soluble Vascular Endothelial Growth Factor Type 2 Receptors (sVEGFR2)
Description: Plasma concentrations of potential pharmacodynamic markers; Soluble Vascular Endothelial Growth Factor Type 2 Receptors (sVEGFR2)
Time Frame: Days 1, 14 and 28 of Cycle 1; Days 1 and 28 of Cycle 2; Day 28 of Cycle 3
Population: as for outcome 15
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Overall
Number analyzed (Participants) | 51
pg/mL
  Cycle 1 Day 1 (n=51) | 9311.00 (1630.73) [5544.00 to 11975.00]
  Cycle 1 Day 14 (n=42) | 4673.50 (1402.34) [2647.00 to 8610.00]
  Cycle 1 Day 28 (n=16) | 3650.00 (1442.21) [2573.00 to 6959.00]
  Cycle 2 Day 1 (n=18) | 7276.50 (1756.36) [4226.00 to 9253.00]
  Cycle 2 Day 28 (n=8) | 3535.00 (927.90) [3093.00 to 5337.00]
  Cycle 3 Day 28 (n=6) | 3312.50 (831.61) [1952.00 to 4742.00]

ADVERSE EVENTS:
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 28/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=51)
Anaemia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Thyroiditis (Endocrine disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Malaise (General disorders) | 2
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 5
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=51)
Anaemia (Blood and lymphatic system disorders) | 15
Palpitations (Cardiac disorders) | 5
Hypothyroidism (Endocrine disorders) | 23
Conjunctivitis (Eye disorders) | 4
Erythema of eyelid (Eye disorders) | 3
Eyelid oedema (Eye disorders) | 13
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 6
Anal erosion (Gastrointestinal disorders) | 4
Cheilitis (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 29
Dyspepsia (Gastrointestinal disorders) | 12
Gastritis (Gastrointestinal disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 3
Gingival swelling (Gastrointestinal disorders) | 3
Gingivitis (Gastrointestinal disorders) | 7
Glossitis (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 5
Lip dry (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 3
Mouth haemorrhage (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 25
Periodontitis (Gastrointestinal disorders) | 3
Periproctitis (Gastrointestinal disorders) | 6
Stomach discomfort (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 26
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 15
Chest pain (General disorders) | 3
Chills (General disorders) | 5
Face oedema (General disorders) | 24
Fatigue (General disorders) | 34
Malaise (General disorders) | 19
Oedema (General disorders) | 8
Oedema peripheral (General disorders) | 21
Pyrexia (General disorders) | 30
Thirst (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 24
Pharyngitis (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 26
Aspartate aminotransferase increased (Investigations) | 35
Blood albumin decreased (Investigations) | 18
Blood alkaline phosphatase increased (Investigations) | 18
Blood amylase increased (Investigations) | 26
Blood bilirubin increased (Investigations) | 16
Blood calcium decreased (Investigations) | 12
Blood creatine phosphokinase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 29
Blood glucose increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 36
Blood phosphorus decreased (Investigations) | 14
Blood potassium increased (Investigations) | 3
Blood pressure increased (Investigations) | 4
Blood sodium decreased (Investigations) | 5
Blood thyroid stimulating hormone increased (Investigations) | 7
Blood urea increased (Investigations) | 8
Blood uric acid increased (Investigations) | 8
Blood urine present (Investigations) | 4
C-reactive protein increased (Investigations) | 10
Gamma-glutamyltransferase increased (Investigations) | 7
Haemoglobin decreased (Investigations) | 25
Lipase increased (Investigations) | 36
Lymphocyte count decreased (Investigations) | 36
Neutrophil count decreased (Investigations) | 41
Platelet count decreased (Investigations) | 47
Protein total decreased (Investigations) | 11
Red blood cell count decreased (Investigations) | 3
Weight decreased (Investigations) | 9
Weight increased (Investigations) | 6
White blood cell count decreased (Investigations) | 44
Anorexia (Metabolism and nutrition disorders) | 36
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Hypoproteinaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 28
Headache (Nervous system disorders) | 13
Hypoaesthesia (Nervous system disorders) | 4
Hypogeusia (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 6
Chromaturia (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 9
Scrotal ulcer (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Achromotrichia acquired (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 8
Eczema (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 8
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 27
Pruritus (Skin and subcutaneous tissue disorders) | 6
Purpura (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 29
Skin discolouration (Skin and subcutaneous tissue disorders) | 37
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin reaction (Skin and subcutaneous tissue disorders) | 7
Yellow skin (Skin and subcutaneous tissue disorders) | 5
Haemorrhage (Vascular disorders) | 3
Hypertension (Vascular disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.